CLINICAL TRIAL: NCT01579227
Title: Efficacy Of Tocotrienol a Natural Vitamin E In Biopsy Wound.
Acronym: TOP/OTOP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chandan K Sen (Other)
Collaborators: Carotech Inc. (Industry)
Responsible Party: Sponsor-Investigator, Chandan K Sen, Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2011H0286
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2017-01

CONDITIONS: Scar
Keywords: Healthy participants
MeSH Terms: conditions — Cicatrix | interventions — Tocotrienols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue biopsy will be collected twice in the study period.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1-TOP group 1: TOP group 1 will have biopsy #2 collected 3 days after 1st biopsy collected.
- TOP group 2: TOP group 2 will have biopsy #2 collected 30 days after 1st biopsy collected.
- OTOP group-1: OTOP will use topical cream (either topical tocotrienol (TCT) or placebo cream) as well as oral supplementation (either oral Tocotrienol capsules (TCT) or placebo capsules). OTOP group 1 will have biopsy #2 collected 3 days after 1st biopsy collected.
  Interventions: Device: Topical Tocotrienol (TCT); Dietary Supplement: Oral Tocotrienol Capsules (TCT); Device: Placebo cream; Dietary Supplement: placebo capsule
- OTOP group-2: OTOP will use topical cream (either topical tocotrienol (TCT) or placebo cream) as well as oral supplementation (either oral Tocotrienol capsules (TCT) or placebo capsules). OTOP group 2 will have biopsy #2 collected 30 days after 1st biopsy collected.
  Interventions: Device: Topical Tocotrienol (TCT); Dietary Supplement: Oral Tocotrienol Capsules (TCT); Device: Placebo cream; Dietary Supplement: placebo capsule
- TAM Group 1: TAM group 1 will have #2 biopsy collected 21 days after 1st biopsy collected. Tamoxifen cream and placebo cream will be applied where biopsies are collected from 1 week prior to having the biopsy procedure until the second biopsy is collected (21 days later).
  Interventions: Device: Tamoxifen Cream
- Normal Skin: Placebo group will apply placebo and TCT cream that will be applied daily to a specified area on the subjects legs (normal skin) for 5 weeks. One leg will be applied with placebo and the other will be applied with TCT cream. Subjects will return weekly for 5 weeks, where non-invasive measurements using Laser Speckle imaging, will be completed at each study visit
  Interventions: Device: Tamoxifen Cream; Device: Placebo cream

INTERVENTIONS:
Device: Topical Tocotrienol (TCT) — Natural Form Vitamin E topical cream(TCT)
  Other Names: TCT
  Groups: OTOP group-1; OTOP group-2
Dietary Supplement: Oral Tocotrienol Capsules (TCT) — Natural Form Vitamin E Oral capsules (TCT)
  Other Names: TCT
  Groups: OTOP group-1; OTOP group-2
Device: Tamoxifen Cream — Tamoxifen cream
  Groups: Normal Skin; TAM Group 1
Device: Placebo cream — Placebo cream
  Other Names: Placebo
  Groups: Normal Skin; OTOP group-1; OTOP group-2
Dietary Supplement: placebo capsule — placebo capsule
  Other Names: placebo
  Groups: OTOP group-1; OTOP group-2

SUMMARY:
The following two objectives are proposed in healthy subjects to characterize (1) wound closure, (2) scar formation/appearance, and (3) inflammatory response:

Objective 1, (topical only - referred to as "TOP") - Topical application of Tocotrienol (TCT) vs placebo in bilateral punch biopsy

Objective 2, (oral and topical - referred to as "OTOP") - Combined oral supplementation and topical application of tocotrienol (TCT) vs placebo in bilateral punch biopsy

Objective 3, (topical only - referred to as "TAM") - Topical application of tamoxifen vs placebo in bilateral punch biopsy.

Objective 4, (topical only to normal skin) - Topical application of TCT vs placebo on bilateral lets on normal skin.

DETAILED DESCRIPTION:
* In nature, the vitamin E family is split into two classes: tocopherols (TCP) and tocotrienols (TCT). Members of the TCP and TCT family are biologically unique.

  * TCP are mainly found in green leafy vegetables while TCT are the primary vitamin E of seeds, including cereal grains such as wheat, rice, and barley.
* Vitamin E is thought to improve wound healing by inhibiting collagen synthesis and attenuating fibroblast proliferation and inflammation. However, outcomes based scientific literature on the therapeutic efficacy of vitamin E in skin wound closure is scant and has primarily focused on TCP.

  * Oral supplementation of TCP showed modest improvement in rodent wound closure, but the relevance of oral TCP supplementation in rats already receiving high dose vitamin E in a standard laboratory is questionable.
  * Topical TCP on surgical wounds of children have been shown to improve wound healing; yet no mechanistic basis for the observed effect was described.
* Preliminary observations from the PI's active IRB protocol to test TCT in scar appearance of surgical wounds led us to evaluate the potential of TCT vitamin E to improve wound closure in healthy subjects. To date, the therapeutic efficacy of TCT in either topical (TOP) or oral with topical (OTOP) applications for skin wound healing remains to be reported.

  * Preliminary observations also made show down-regulation of microRNA-200b supports cutaneous angiogenesis, the most important step in cutaneous wound healing. Tamoxifen silences mircroRNA-200b and later work has recognized that under non-neoplastic conditions, tamoxifen may induce angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Ages- 18-50 (Both Male & Female)
* Non-smoker - having quit at least 3 months prior to enrollment
* Non-diabetic
* Non-pregnant or non-breastfeeding - verbal assent.
* If a female subject of childbearing age misses her menstrual period after the start of the study, she will inform the investigators and be given a pregnancy test to ensure, for safety reasons, that she is not pregnant. If she is pregnant, she will discontinue participation in the study.
* No current use of OTC medications or other form of supplements containing vitamin-E

Exclusion Criteria:

* Diabetes or HIV diagnosis
* Alcohol or drug abuse
* unable to provide informed consent
* Therapeutically anti-coagulated
* Prisoner
* Currently prescribed immunosuppressant medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We plan to recruit 27 healthy adult subjects for the TOP group, 34 healthy adult subjects for the OTOP group,10 healthy adult subjects for the TAM group and 30 healthy subjects for Normal Skin.
Sampling Method: Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2012-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
WOUND CLOSURE | 1-2 month(s)
  Wound closure will be assessed by results of conventional camera and thermal imaging in Group 1 and Group 2 subjects.

SECONDARY OUTCOMES:
SCARRING | 1-2 month (s)
  Scarring will be assessed in group 1 and group 2 subjects by the Vancouver Scar Scale (VSS). Scoring will be performed by three blinded observers. The VSS evaluates vascularity (redness), height (hypertrophy), pliability (contracture and elastic texture) and pigmentation.

OTHER OUTCOMES:
Wound closure and Increased Angiogenesis | 1-2 months
  Test whether miR-200b is silenced with tamoxifen resulting in increased angiogenesis and faster wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States